CLINICAL TRIAL: NCT01728220
Title: A Placebo-Controlled, Double-Blind, Parallel, Randomized, Two-Part, Clinical Dose-Confirming Study Of Pulsed, Inhaled Nitric Oxide (iNO) In Subjects With World Health Organization (WHO) Group 3 Pulmonary Hypertension (PH) Associated With Chronic Obstructive Pulmonary Disease (COPD) On Long Term Oxygen Therapy (LTOT) INHALE 1
Brief Title: Two-Part Dose-Confirming Study of Pulsed Inhaled Nitric Oxide in Subjects With WHO Group 3 Pulmonary Hypertension Associated With COPD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bellerophon Pulse Technologies (Industry)
Responsible Party: Sponsor
Organization: Bellerophon (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IK-7002-COPD-201
Record Dates: First submitted 2012-11-13; First posted 2012-11-19 (Estimated); Last update posted 2023-02-27 (Actual); Status verified 2022-07

CONDITIONS: Pulmonary Hypertension; Chronic Obstructive Pulmonary Disease
Keywords: Inhaled nitric oxide (iNO); Pulmonary hypertension (PH); Chronic obstructive pulmonary disease (COPD); Long term oxygen therapy (LTOT)
MeSH Terms: conditions — Hypertension, Pulmonary; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (7):
- Inhaled NO @ 0.003 mg/kg/ ideal body weight (IBW)/hr (Part A) (Active Comparator): Inhaled NO using 3.0 mg/L [2440 ppm] NO minicylinder delivered via INOpulse® DS-C device
  Interventions: Combination Product: Inhaled NO delivered via INOpulse DS-C Device
- Inhaled NO @ 0.010 mg/kg/IBW/hr (Part A) (Active Comparator): Inhaled NO using 3.0 mg/L [2440 ppm] NO minicylinder delivered via INOpulse® DS-C device
  Interventions: Combination Product: Inhaled NO delivered via INOpulse DS-C Device
- Inhaled NO @ 0.015 mg/kg/IBW/hr (Part A) (Active Comparator): Inhaled NO using 6.0 mg/L [4880 ppm] NO minicylinder delivered via INOpulse® DS-C device
  Interventions: Combination Product: Inhaled NO delivered via INOpulse DS-C Device
- Placebo random @ 0.003, 0.010 or 0.015 mg/kg/IBW/hr (Part A) (Placebo Comparator): Placebo using 99.999% N2 minicylinder delivered via INOpulse® DS-C device
  Interventions: Combination Product: Placebo delivered via INOpulse DS-C Device
- Inhaled NO @ 0.030 mg/kg IBW/hr (Part B) (Active Comparator): Inhaled NO using 6.0 mg/L [4880 ppm] NO minicylinder delivered via INOpulse® DS-C device
  Interventions: Combination Product: Inhaled NO delivered via INOpulse DS-C Device
- Inhaled NO @ 0.075 mg/kg IBW/hr (Part B) (Active Comparator): Inhaled NO using 6.0 mg/L [4880 ppm] NO minicylinder delivered via INOpulse® DS-C device
  Interventions: Combination Product: Inhaled NO delivered via INOpulse DS-C Device
- Placebo random @ 0.030 or 0.075 mg/kg/IBW (Part B) (Active Comparator): Placebo using 99.999% N2 minicylinder delivered via INOpulse® DS-C device
  Interventions: Combination Product: Placebo delivered via INOpulse DS-C Device

INTERVENTIONS:
Combination Product: Inhaled NO delivered via INOpulse DS-C Device — Subjects will be treated with nitric oxide by means of an INOpulse DS-C device using an INOpulse nasal cannula.
  Arms: Inhaled NO @ 0.003 mg/kg/ ideal body weight (IBW)/hr (Part A); Inhaled NO @ 0.010 mg/kg/IBW/hr (Part A); Inhaled NO @ 0.015 mg/kg/IBW/hr (Part A); Inhaled NO @ 0.030 mg/kg IBW/hr (Part B); Inhaled NO @ 0.075 mg/kg IBW/hr (Part B)
Combination Product: Placebo delivered via INOpulse DS-C Device — Subjects will be treated with nitrogen gas by means of an INOpulse DS-C device using an INOpulse nasal cannula.
  Arms: Placebo random @ 0.003, 0.010 or 0.015 mg/kg/IBW/hr (Part A); Placebo random @ 0.030 or 0.075 mg/kg/IBW (Part B)

SUMMARY:
This is a placebo-controlled, double-blind, parallel, randomized, two-part, dose-confirming clinical study characterizing the pharmacodynamic effects of pulsed iNO using the combination product, inhaled nitric oxide/INOpulse DS-C vs. placebo in subjects with World Health Organization (WHO) Group 3 pulmonary hypertension (PH) associated with Chronic Obstructive Pulmonary Disease (COPD) on Long Term Oxygen Therapy (LTOT).

DETAILED DESCRIPTION:
This two-part study is designed to confirm the dose of inhaled nitric oxide (NO), administered through an investigational pulsed delivery device (INOpulse® DS-C) that results in decreased pulmonary arterial systolic pressure (PASP) without significantly affecting systemic oxygenation.

In Part A, 80 subjects will be randomized to 1of 4 treatment groups in a 1:1:1:1 ratio (with 20 subjects in each treatment group). Subjects assigned to an iNO group will receive pulsed iNO at a dose of 0.003 mg/kg IBW/hr, 0.010 mg/kg IBW/hr, or 0.015 mg/kg IBW/hr, with a set pulse width (PW) of 260 milliseconds (ms). Part A subjects assigned to the placebo group will receive nitrogen (N2) at a randomly assigned device setting of 0.003, 0.010 or 0.015 mg/kg IBW/hr with a set PW of 260 ms.

Subjects who were randomized in Part A are permitted to participate in Part B of the study. Subjects will need to be re-screened and re-randomized for Part B participation.

In Part B, 60 subjects will be randomized to 1 of 3 treatment groups in a 1:1:1 ratio (with 20 subjects in each treatment group). Subjects assigned to an iNO group will receive pulsed iNO at either 0.030 mg/kg IBW/hr or 0.075 mg/kg IBW/hr, with a set PW of 260 ms. Part B subjects assigned to placebo will receive N2 at a randomly assigned device setting of 0.030 mg/kg IBW/hr or 0.075 mg/kg IBW/hr with a set PW of 260 ms.

Part B will use a skewed block randomization scheme with 10 blocks of 6 subjects as follows:

* Blocks 1-3: 3 subjects at 0.030 mg/kg IBW/hr, 1 subject at 0.075 mg/kg IBW/hr, and 2 subjects randomly assigned to placebo either 0.030 or 0.075 mg/kg IBW/hr
* Blocks 4-7: 2 subjects at 0.030 mg/kg IBW/hr, 2 subjects at 0.075 mg/kg IBW/hr, and 2 subjects randomly assigned to placebo either 0.030 or 0.075 mg/kg IBW/hr
* Blocks 8-10: 1 subject at 0.030 mg/kg IBW/hr, 3 subjects at 0.075 mg/kg IBW/hr, and 2 subjects randomly assigned to placebo either 0.030 or 0.075 mg/kg IBW/hr

ELIGIBILITY:
Inclusion Criteria:

1. Former smokers with at least 10 pack-years of tobacco cigarette smoking history before study entry and who have stopped smoking ≥ 1 month prior to enrollment
2. Age ≥ 40 years, ≤ 80 years
3. A confirmed diagnosis of COPD by the Global initiative for chronic Obstructive Lung Disease (GOLD) criteria
4. A post-bronchodilatory forced expiratory volume in 1 second/forced vital capacity (FEV1/FVC) < 0.7 and a FEV1 < 60% predicted (values obtained within 6 months prior to screening can be used unless obtained within ± 7 days of an exacerbation; otherwise, the test must be performed during screening)
5. Receiving LTOT for ≥ 3 months and ≥ 10 hours per day as determined by history
6. Echocardiogram with technical adequacy demonstrating tricuspid regurgitation velocity (TRV) ≥ 2.9 m/s at Screening, as determined by a blinded central echocardiography laboratory
7. Females of childbearing potential must have a negative pre-treatment urine pregnancy test
8. Signed informed consent prior to the initiation of any study mandated procedures or assessments

Exclusion criteria:

Subjects who meet any of the following criteria are not eligible for enrollment:

1. Positive urine cotinine test
2. Currently using, or having used within the past month, a nicotine patch
3. A diagnosis of asthma or other non-COPD respiratory disease, in the opinion of the Investigator
4. Lack of patency of nares upon physical examination
5. Experienced an exacerbation requiring start of or increase in systemic oral corticosteroid therapy and/or hospitalization during the last month (ATS COPD Guidelines 2004)
6. Left ventricular dysfunction as measured by:

   1. Screening echocardiographic evidence of left ventricular systolic dysfunction (left ventricular ejection fraction (LVEF) < 40%), or
   2. Screening echocardiographic evidence of left ventricular diastolic dysfunction > moderate (i.e., > Grade 2), or
   3. Any history of pulmonary capillary wedge pressure (PCWP), left atrial pressure (LAP) or left ventricular end diastolic pressure (LVEDP) > 18 mm Hg as measured during cardiac catheterization within the past 6 months unless documented to have resolved by a subsequent cardiac catheterization
7. Clinically significant valvular heart disease that may contribute to PH, including mild or greater aortic valvular disease (aortic stenosis or regurgitation) and/or moderate or greater mitral valve disease (mitral stenosis or regurgitation), or status post mitral valve replacement
8. Use within 30 days of screening or current use of approved PH medications such as sildenafil or bosentan (use of Cialis® or Viagra® for erectile dysfunction is permitted)
9. Use of investigational drugs or devices within 30 days prior to enrollment into the study
10. Any underlying medical or psychiatric condition that, in the opinion of the Investigator, makes the subject an unsuitable candidate for the study

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 159 (Actual)
Dates: Start 2012-12; Primary Completion 2014-06 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Change in pulmonary arterial systolic pressure (PASP) from Baseline after treatment with iNO (measured by 2D transthoracic echocardiography with Doppler) | baseline to end of treatment (1 day)

SECONDARY OUTCOMES:
The secondary outcome is the occurrence of a decrease ≥ 5 mm Hg of partial pressure of oxygen in arterial blood (PaO2) from Baseline after treatment with iNO | baseline to end of treatment (1 day)

CONTACTS AND LOCATIONS:
Overall Officials: Ashika Ahmed, MD, Study Director — Bellerophon Therapeutics
Locations (43):
- United States (43):
  - Jasper Summit Research LLC, Jasper, Alabama
  - Clinical Trial Connection, Flagstaff, Arizona
  - Pulmonary Associates P.A., Phoenix, Arizona
  - Radin Cardiovascular Medical Associates, Newport Beach, California
  - Western Connecticut Medical Group PC, Danbury, Connecticut
  - Waterbury Pulmonary Associates, Waterbury, Connecticut
  - Bay Area Chest Physicians, Clearwater, Florida
  - Gary J. Richmond, MD, PA, Fort Lauderdale, Florida
  - East Coast Institute for Research, Jacksonville, Florida
  - Pulmonary Disease Specialists PA, Kissimmee, Florida
  - San Marcus Research Clinic Inc., Miami, Florida
  - St. Paul Medical Research Center Inc., Miami, Florida
  - IMIC, Inc., Miami, Florida
  - Elite Clinical Research, Miami, Florida
  - South Florida Research Phase I-IV, Miami, Florida
  - Health & Life Research Solutions Inc., Miami, Florida
  - Advanced Research Institute, Inc., New Port Richey, Florida
  - Central Florida Pulmonary Group, P.A., Orlando, Florida
  - Bassette Medical Research Inc., Sebring, Florida
  - Research Alliance, St. Petersburg, Florida
  - Concept Clinical Trials, LLC, Tamarac, Florida
  - Axcess Medical Research, Wellington, Florida
  - Florida Premier Research Institute, Winter Park, Florida
  - River Birch Research Alliance LLC, Blue Ridge, Georgia
  - Medical Associates of North Georgia, Canton, Georgia
  - Veritas Clinical Specialties, Ltd, Topeka, Kansas
  - Graves-Gilbert Clinic, Bowling Green, Kentucky
  - Kentucky Research Group, Louisville, Kentucky
  - MedPharmics LLC, Metairie, Louisiana
  - Physician HealthCare Network, PC, Port Huron, Michigan
  - Montefiore Medical Center-Weiler Division, The Bronx, New York
  - American Health Research, Charlotte, North Carolina
  - University Hospitals Case Medical Center, Cleveland, Ohio
  - Temple Lung Center Pulmonary & Critical Care Medicine, Philadelphia, Pennsylvania
  - Lowcountry Lung and Critical Care, Charleston, South Carolina
  - Neem Research Group Inc, Columbia, South Carolina
  - Gaffney Pharmaceutical Research, Gaffney, South Carolina
  - Greenville Pharmaceutical Research, Greenville, South Carolina
  - Clinical Research of Rock Hill, Rock Hill, South Carolina
  - Spartanburg Medical Research, Spartanburg, South Carolina
  - Pioneer Research Solutions, Inc., Sugar Land, Texas
  - Pulmonary Associates of Richmond Inc, Richmond, Virginia
  - Zain Research LLC, Richland, Washington